CLINICAL TRIAL: NCT04134520
Title: PL-210: Establish ProLung Test Measurement Collection Protocol for Future Studies.
Brief Title: Establish ProLung Test Measurement Collection Protocol for Future Studies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fresh Medical Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: PL 210
Record Dates: First submitted 2019-10-09; First posted 2019-10-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Cancer , Healthy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Generally healthy subjects with no known cancer disorder
  Interventions: Device: ProLung System
- Subjects with a pathological diagnosis of cancer
  Interventions: Device: ProLung System

INTERVENTIONS:
Device: ProLung System — Non-invasive bioconductance measurements

SUMMARY:
The purpose of this Study is to identify and test different data collection methods to determine which approaches improve the ProLung Testing procedure. Once this Study is complete, the Sponsor plans to evaluate these improvements in future follow up Validation studies that will assess device accuracy using the new measurement collection methods.

ELIGIBILITY:
Inclusion Criteria:

7 2.0 Study Objectives 2.1 Objectives and Aims The purpose of this Study is to identify and test different data collection methods to determine which approaches improve the ProLung Testing procedure and identify approaches that may be useful in evaluating other cancers in addition to lung cancer. Once this Study is complete, the Sponsor plans to evaluate these improvements in future follow up cancer validation studies that will assess device accuracy using the new measurement collection methods.

The Specific Aim of this study:

1. Establish the ProLung Test measurement collection protocol for future studies.
2. Assess the safety and tolerability of the ProLung Test procedures. 3.0 Study Design This Study Non-Interventional Observational Multi-Site Study in which the ProLung Test does not affect, influence or alter the subject's normal standard of care. The Study will collect data from multiple sites (1- 15). The Study will enroll a minimum of 100 and a maximum 500 subjects. Each subject will receive one or multiple measurement sessions on separate days. 3.1 Safety and Tolerability Information collected about adverse events and tolerability will be analyzed as described in sections 5.8 and 6.0 (Additional Data Collection and Adverse Events). 3.2 Monitoring The study Sponsor will provide monitors to monitor Protocol compliance and provide guidance pertaining to the management of the Study. 4.0 Subject Selection and Participation 4.1 Inclusion Criteria

Subjects who meet all of the following criteria may be enrolled in this Study:

1. Subject is male or female, age 18 or older.
2. Subjects eligible for enrollment in one of three arms as described herein Arm 1: Generally healthy subjects with no known cancer disorder Arm 2: Subjects with a pathological diagnosis of cancer that have not yet received treatment for cancer Arm 3: Subjects with a finding that is suspicious for cancer and have not been pathologically confirmed for cancer and have not yet received treatment for cancer Arm 4: Subjects with a cancer finding that has been pathologically confirmed as benign
3. Subject is capable of understanding and agreeing to fulfill the requirements of this Protocol.
4. Subject has signed the IRB/IEC approved Informed Consent Form ("ICF").

Exclusion Criteria:

The following criteria will disqualify a subject from enrollment into this Study:

1. Subject has an implanted electronic device in the chest.
2. Subject presents with an anomalous physical or anatomical condition that precludes ProLung Test measurement.
3. Subject will have undergone unusually strenuous exercise within 24 hours.
4. Subject who has significant systemic diseases such as uncontrolled diabetes, advanced heart failure, or a recent myocardial infarction, or other medical condition such as severe morbid obesity that in the judgment of the Principal Investigator would make him/her unsuitable for the Study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Arm 1: Generally healthy subjects with no known cancer disorder Arm 2: Subjects with a pathological diagnosis of cancer that have not yet received treatment for cancer Arm 3: Subjects with a finding that is suspicious for cancer and have not been pathologically confirmed for cancer and have not yet received treatment for cancer Arm 4: Subjects with a cancer finding that has been pathologically confirmed as benign
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-10-16 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Establish the ProLung Test measurement collection protocol for future studies. | 1 day
  The study will evaluate several data collection methodologies including the China CFDA Study method which utilizes diaphoretic electrodes as the reference electrode at measurement point locations and other methods using brass reference electrode at point locations. In addition, the benefits of obtaining multiple repeat measurements will be evaluated.

SECONDARY OUTCOMES:
Assess the safety and tolerability of the ProLung Test procedures | 1 day
  Adverse events will be recorded and following the ProLung Test, subjects will be asked to complete a brief questionnaire regarding their experience and perception of the procedure. The questions are:
  1. Did the test cause any discomfort? If so, please describe.
  2. Did the time required for measurement seem too long? If so, what amount of time seems reasonable?
  3. Would you undergo measurement again? If so, please describe
  4. Do you have any suggestions for improving the measurement procedure? If so, please describe.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Coastal Pulmonary Associates, Encinitas, California
  - Loyola Medical University, Maywood, Illinois
  - Ogden Regional Medical Center, Ogden, Utah
  - Michael Garff, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No